CLINICAL TRIAL: NCT05571137
Title: A Multinational, Non-Interventional, Retrospective Study on CMV Infection Outcomes, Treatment Patterns and Healthcare Utilization Study (OTUS) Among Hematopoietic Stem Cell Transplant (HSCT) Recipients in Europe and Canada (OTUS HSCT Extension in the EUCAN Countries: Austria, Belgium, Canada, Greece, Israel, Netherlands, Poland and Serbia)
Brief Title: A Study on Cytomegalovirus (CMV) Infection Outcomes Among Hematopoietic Stem Cell Transplant (HSCT) Participants in Europe and Canada
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-620-4004
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Cytomegalovirus (CMV)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Resistant, Refractory, or Intolerant (RRI) to Anti-CMV treatment: Participants who had a HSCT after January 1, 2016, and developed post-transplant CMV infection were subsequently characterized as RRI to currently available anti-CMV treatment for at least 12 months before being enrolled, will be observed in this retrospective study for 24 months.
- Cohort 2: Pre-emptive CMV Treatment: Participants who had a HSCT after January 1, 2019, were preemptively treated for CMV for at least 12 months before being enrolled, will be observed in this retrospective study for 24 months.

SUMMARY:
The main aim of the study is to assess the clinical outcomes of current CMV management across different regions of the world (Europe [EU] and Canada [CAN]). Data will be collected retrospectively from medical charts.

No study medicines will be provided to participants in this study.

DETAILED DESCRIPTION:
This study consists of two cohorts: Cohort 1 (resistant, refractory or intolerant to anti-CMV agents) includes participants who had an HSCT after January 1, 2016. Cohort 2 (pre-emptive treatment for CMV viremia) includes participants who had an HSCT after January 1, 2019. Participants who meet the criteria for both cohorts will be evaluated in each cohort separately (i.e., Cohort 1 and Cohort 2 are not mutually exclusive, and participants will be analyzed in both cohorts using unique index dates with respect to the cohort-specific eligibility criteria). Participant follow-up in the medical record must be available for at least one year from the CMV index date or death, whichever occurs first. The start date of data collection corresponds to the end of participant follow up. For Cohort 1, it is expected that follow up data will be available for up to 7 years (for those participants with an index date in 2016 and followed through 2022). For Cohort 2, it is expected that follow-up data will be available for up to 4 years (for those participants with an index date in 2019 and followed through 2022).

ELIGIBILITY:
Inclusion Criteria:

(Cohort 1) Resistant / Refractory or Intolerant:

* Aged greater than and equal to (>=) 18 years at the time of the HSCT.
* Received an HSCT after January 1, 2016.
* Diagnosed with CMV infection any time after the HSCT date.
* Required >=1 anti-CMV agent to manage CMV infection and were subsequently considered:

  1. resistant to currently available anti-CMV agent; OR
  2. refractory to currently available anti-CMV agent; OR
  3. intolerant to currently available anti-CMV agent.
* Follow-up information is available for at least 12 months from the index date (i.e., date when the participant was first considered resistant, refractory or intolerant to anti-CMV agent) or death, whichever occurs first.
* Provided written informed consent prior to the initiation of any study procedures (unless waiver was granted by Institutional Ethical Committee [IEC]).

(Cohort 2) Pre-emptive treatment for CMV viremia:

* Aged >=18 years at the time of the HSCT.
* Received an HSCT after January 1, 2019.
* Diagnosed with CMV viremia any time after the HSCT date and received pre-emptive anti-CMV agent.
* Follow-up information is available for at least 12 months from the index date (i.e., date when the patient was first preemptively treated with an anti-CMV agent) or death, whichever occurs first.
* Provided written informed consent prior to the initiation of any study procedures (unless waiver was granted by IEC).

Exclusion Criteria (both cohorts)

* Diagnosed as being positive for human immunodeficiency virus before the HSCT.
* Unable to demonstrate a minimum of 12 months of follow-up from the index date (e.g., incomplete information on dates showing follow-up time).
* Participation in a clinical trial related to CMV treatment during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who had a CMV infection treated with at least one anti-CMV agent and considered resistant, refractory, or intolerant to a currently available agent will be enrolled in Cohort 1 and participants who received pre-emptive therapy for CMV viremia will be enrolled in Cohort 2.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Time From HSCT Until Start of Asymptomatic and Symptomatic Index Episode | From HSCT up to start date of the index episode (Up to 7 years 3 months)
  Index episode is first CMV episode in which the participant is considered RRI to anti-CMV treatment or had CMV viremia and received pre-emptive treatment, without becoming RRI during that episode. Symptomatic episode is an episode wherein there is "Tissue invasive/end organ disease" or "CMV syndrome" at any time, and asymptomatic when there is no such observation.
Percentage of Participants who are Asymptomatic and Symptomatic at the Index and Recurrent Episodes | Up to 7 years 3 months
  Index episode is first CMV episode in which the participant is considered RRI to anti-CMV treatment or had CMV viremia and received pre-emptive treatment, without becoming RRI during that episode. Recurrent episodes are defined as new CMV infection in a participant with previous evidence of CMV infection. Symptomatic episode is an episode wherein there is "tissue invasive/end organ disease" or "CMV syndrome" at any time, and asymptomatic when there is no such observation.
Percentage of Participants With CMV Viremia Clearance as Defined by Site Investigator at the Index and Recurrent Episodes | Up to 7 years 3 months
  Index episode is first CMV episode in which the participant is considered RRI to anti-CMV-treatment or had CMV viremia and received pre-emptive treatment, without becoming RRI during that episode. Recurrent episodes is defined as new CMV infection in a participant with previous evidence of CMV infection. CMV viremia clearance is defined as when an active CMV viremia can be considered cleared from the participant, as determined by the site investigator.
Time From Start of Index Episode to CMV Viremia Clearance as Defined by Site Investigator | From start of index episode to CMV viremia clearance (Up to 7 years 3 months)
  Index episode is first CMV episode in which the participant is considered RRI to anti-CMV treatment or had CMV viremia and received pre-emptive treatment, without becoming RRI during that episode. CMV viremia clearance is defined as when an active CMV viremia can be considered cleared from the participant, as determined by the site investigator.
Percentage of Participants With CMV Viremia Clearance as Defined by Site Investigator at Week 8 After Index Date | At Week 8 after index date
  Index date is the date when participant was considered resistant, refractory or intolerant to anti-CMV treatment for the first time after transplant (RRI CMV index date) or pre-emptive treatment for the first time after transplant following CMV viremia (CMV preemptive treatment index date). CMV viremia clearance is defined as when an active CMV viremia can be considered cleared from the participant, as determined by the site investigator. The assessment will be based on Kaplan-Meier estimate.
Percentage of Participants With CMV Viremia Clearance as Defined by Site Investigator at Week 20 After Index Date | At Week 20 after index date
  Index date is the date when participant was considered resistant, refractory or intolerant to anti-CMV treatment for the first time after transplant (RRI CMV index date) or pre-emptive treatment for the first time after transplant following CMV viremia (CMV preemptive treatment index date). CMV viremia clearance is defined as when an active CMV viremia can be considered cleared from the participant, as determined by the site investigator. The assessment will be based on Kaplan-Meier estimate.
Percentage of Participants With CMV Viremia Clearance as Defined by Site Investigator at 1-year After Index Date | At 1-year after index date
  Index date is the date when participant was considered resistant, refractory or intolerant to anti-CMV treatment for the first time after transplant (RRI CMV index date) or pre-emptive treatment for the first time after transplant following CMV viremia (CMV preemptive treatment index date). CMV viremia clearance is defined as when an active CMV viremia can be considered cleared from the participant, as determined by the site investigator. The assessment will be based on Kaplan-Meier estimate.
Percentage of Participants With Non-Detectable CMV During the Index Episode Prior to and After the Index Date | Up to 7 years 3 months
  Index episode is first CMV episode in which the participant is considered RRI to anti-CMV treatment or had CMV viremia and received pre-emptive treatment, without becoming RRI during that episode. Index date is the date when participant was considered resistant, refractory or intolerant to anti-CMV treatment for the first time after transplant (RRI CMV index date) OR pre-emptive treatment for the first time after transplant following CMV viremia (CMV preemptive treatment index date). Non-detectable CMV is defined as highest minimum detectable level of CMV assays across all transplant sites.
Percentage of Participants With Non-Detectable CMV at Week 8 After Index Date | At Week 8 after index date
  Index date is the date when participant was considered resistant, refractory or intolerant to anti-CMV treatment for the first time after transplant (RRI CMV index date) or pre-emptive treatment for the first time after transplant following CMV viremia (CMV preemptive treatment index date). Non-detectable CMV is defined as highest minimum detectable level of CMV assays across all transplant sites. The assessment will be based on Kaplan-Meier estimate.
Percentage of Participants With Non-Detectable CMV at Week 20 After Index Date | At Week 20 after index date
  Index date is the date when participant was considered resistant, refractory or intolerant to anti-CMV treatment for the first time after transplant (RRI CMV index date) or pre-emptive treatment for the first time after transplant following CMV viremia (CMV preemptive treatment index date). Non-detectable CMV is defined as highest minimum detectable level of CMV assays across all transplant sites. The assessment will be based on Kaplan-Meier estimate.
Percentage of Participants With Non-Detectable CMV at 1-year After Index Date | At 1-year after index date
  Index date is the date when participant was considered resistant, refractory or intolerant to anti-CMV treatment for the first time after transplant (RRI CMV index date) or pre-emptive treatment for the first time after transplant following CMV viremia (CMV preemptive treatment index date). Non-detectable CMV is defined as highest minimum detectable level of CMV assays across all transplant sites. The assessment will be based on Kaplan-Meier estimate.
Time From Treatment Initiation to CMV Viremia Clearance as Defined by Site Investigator at the Index Episode | From Treatment Initiation to CMV Viremia Clearance (Up to 7 years 3 months)
  Index episode is first CMV episode in which the participant is considered RRI to anti-CMV treatment or had CMV viremia and received pre-emptive treatment, without becoming RRI during that episode. CMV viremia clearance is defined as when an active CMV viremia can be considered cleared from the participant, as determined by the site investigator.
Time From Treatment Initiation Until Evidence of Non-detectable CMV at the Index Episode | Time from treatment initiation until evidence of non-detectable CMV (Up to 7 years 3 months)
  Index episode is first CMV episode in which the participant is considered RRI to anti-CMV treatment or had CMV viremia and received pre-emptive treatment, without becoming RRI during that episode. Non-detectable CMV is defined as highest minimum detectable level of CMV assays across all transplant sites.
Time From Start of Index Episode to First Symptomatic CMV Diagnosis | From start of index episode to first symptomatic CMV diagnosis (Up to 7 years 3 months)
  Index episode is first CMV episode in which the participant is considered RRI to anti-CMV treatment or had CMV viremia and received pre-emptive treatment, without becoming RRI during that episode. Symptomatic CMV is defined CMV-related tissue invasive disease or CMV syndrome. Time from start of index episode to first symptomatic CMV diagnosis (tissue invasive disease diagnosis) will be reported.
Time From Stop Date of the Index Episode to First Recurrent Asymptomatic and Symptomatic CMV Viremia | From stop date of the index episode to first recurrent asymptomatic and symptomatic CMV viremia (Up to 7 years 3 months)
  Index episode is first CMV episode in which the participant is considered RRI to anti-CMV treatment or had CMV viremia and received pre-emptive treatment, without becoming RRI during that episode. Recurrent episodes is defined as new CMV infection in a participant with previous evidence of CMV infection.
Percentage of Participants With Anti-CMV Treatment-related Myelosuppression and Nephrotoxicity | Up to 7 years 3 months
  Index episode is first CMV episode in which the participant is considered RRI to anti-CMV treatment or had CMV viremia and received pre-emptive treatment, without becoming RRI during that episode. Percentage of participants with anti-CMV treatment-related myelosuppression and each type nephrotoxicity overall and during the index episode will be reported.
Percentage of Participants With Engraftment From HSCT | Up to 7 years 3 months
  Engraftment is the process by which hematopoietic stem cells (HSC) make their way (homing) to free bone marrow (BM) niches where they can find optimal conditions to survive and proliferate. Percentage of participants with engraftment from HSCT will be reported.
Percentage of Participants With Graft Versus Host Disease (GvHD) From HSCT and Index Date | Up to 7 years 3 months
  Index date is the date when participant was considered resistant, refractory or intolerant to anti-CMV treatment for the first time after transplant (RRI CMV index date) or pre-emptive treatment for the first time after transplant following CMV viremia (CMV preemptive treatment index date. Percentage of participants with GvHD (acute, chronic) from HSCT and from the index date will be reported.
Percentage of Participants With Graft Failure From HSCT and Index Date | Up to 7 years 3 months
  Index date is the date when participant was considered resistant, refractory or intolerant to anti-CMV treatment for the first time after transplant (RRI CMV index date) or pre-emptive treatment for the first time after transplant following CMV viremia (CMV preemptive treatment index date. Graft failure is defined as a serious complication of allogeneic hematopoietic stem cell transplantation (allo-HSCT) defined as either lack of initial engraftment of donor cells (primary graft failure) or loss of donor cells after initial engraftment (secondary graft failure). Percentage of participants with graft failure (primary/secondary) from HSCT and index date will be reported.
Percentage of Participants who Died due to any Cause From HSCT and Index Date | Up to 7 years 3 months
  Index date is the date when participant was considered resistant, refractory or intolerant to anti-CMV treatment for the first time after transplant (RRI CMV index date) or pre-emptive treatment for the first time after transplant following CMV viremia (CMV preemptive treatment index date. Percentage of participants who died due to any cause from HSCT and from the index date will be reported.
Percentage of Participants who Died due to CMV Infection From HSCT and Index Date | Up to 7 years 3 months
  Index date is the date when participant was considered resistant, refractory or intolerant to anti-CMV treatment for the first time after transplant (RRI CMV index date) or pre-emptive treatment for the first time after transplant following CMV viremia (CMV preemptive treatment index date. Percentage of participants who died due to CMV infection from HSCT and the index date will be reported.
Number of Genetic Mutations Conferring Anti-CMV Resistance From HSCT and at Index Episode | Up to 7 years 3 months
  Index episode is first CMV episode in which the participant is considered RRI to anti-CMV treatment or had CMV viremia and received pre-emptive treatment, without becoming RRI during that episode. Genetic mutation includes UL27, UL54, UL56, UL97, other, unknown mutation. Number of genetic mutations conferring anti-CMV resistance from HSCT and at index date will be reported.
Percentage of Participants With a Genetic Mutation Conferring Anti-CMV Resistance From HSCT and at Index Episode | Up to 7 years 3 months
  Index episode is first CMV episode in which the participant is considered RRI to anti-CMV treatment or had CMV viremia and received pre-emptive treatment, without becoming RRI during that episode. Genetic mutation includes UL27, UL54, UL56, UL97, other, unknown mutation. Percentage of participants with a genetic mutation (i.e., UL27, UL54, UL56, UL97, other, unknown) conferring anti-CMV resistance from HSCT and at the index episode will be reported.

SECONDARY OUTCOMES:
Percentage of Participants With Anti-CMV Primary or Secondary Prophylaxis and Pre-emptive Treatment | Up to 7 years 3 months
  Primary Prophylaxis: When the start date of the anti-CMV prophylaxis was prior to start date of first CMV episode. Secondary Prophylaxis: When the start date of the anti-CMV prophylaxis was on/ after the end date of the previous CMV episode and before the start date of the subsequent CMV episode, or if the start date of the anti-CMV was after the last CMV episode. Pre-emptive treatment is defined as anti-CMV treatment was initiated preemptively when the plasma CMV DNA concentration necessitated therapy based on the risk profile of the participant per clinical judgement. Recurrent episodes is defined as new CMV infection in a participant with previous evidence of CMV infection. Index episode is first CMV episode in which the participant is considered RRI to anti-CMV treatment. Percentage of participants with anti-CMV primary or secondary prophylaxis and pre-emptive treatment overall, at the index episode and for recurrent episodes will be reported.
Number of Anti-CMV Therapies Used for Primary or Secondary Prophylaxis and Pre-emptive Treatment | Up to 7 years 3 months
  Primary Prophylaxis is defined as when the start date of the anti-CMV prophylaxis was prior to start date of first CMV episode. Secondary Prophylaxis is defined as when the start date of the anti-CMV prophylaxis was on/ after the end date of the previous CMV episode and before the start date of the subsequent CMV episode, or if the start date of the anti-CMV was after the last CMV episode. Preemptive treatment is defined as anti-CMV treatment was initiated preemptively when the plasma CMV DNA concentration necessitated therapy based on the risk profile of the participant per clinical judgement. Number of anti-CMV therapies used for primary/secondary prophylaxis and pre-emptive treatment will be reported.
Duration of Anti-CMV Prophylaxis Therapy | Up to 7 years 3 months
  Duration of anti-CMV prophylaxis therapy will be reported.
Percentage of Participants With Mono-therapy and Dual-therapy of Anti-CMV Agents of Interest During CMV Episodes | Up to 7 years 3 months
  Monotherapy of anti-CMV agents of interest includes specifically ganciclovir, valganciclovir, foscarnet, cidofovir, letermovir and maribavir, and dual therapy, namely ganciclovir and foscarnet, valganciclovir and foscarnet, cidofovir and valganciclovir, cidofovir and valganciclovir, others which includes acyclovir, valacyclovir, immunoglobulin G (IgG), etc. CMV episode is generally characterized by elevated CMV viremia levels resulting in anti-CMV treatment. Index episode is first CMV episode in which the participant is considered RRI to anti-CMV treatment or had CMV viremia and received pre-emptive treatment, without becoming RRI during that episode. Recurrent episodes is defined as new CMV infection in a participant with previous evidence of CMV infection. Percentage of participants with mono-therapy and dual-therapy of anti-CMV agents of interest during CMV episodes overall, at the index episode and for recurrent episodes will be reported.
Number of Individual and Dual-therapy of Anti-CMV Agents Used During CMV Episodes | Up to 7 years 3 months
  CMV episode is generally characterized by elevated CMV viremia levels resulting in anti-CMV treatment. Index episode is first CMV episode in which the participant is considered RRI to anti-CMV treatment or had CMV viremia and received pre-emptive treatment, without becoming RRI during that episode. Number of individual and dual-therapy of anti-CMV agents used during CMV episodes will be reported.
Number With Individual and Dual Therapy of Anti-CMV Agents Used by Line of Treatment During Index Episode | Up to 7 years 3 months
  Index episode is first CMV episode in which the participant is considered RRI to anti-CMV treatment or had CMV viremia and received pre-emptive treatment, without becoming RRI during that episode. Number of individual and dual therapy of anti-CMV agents used by line of treatment overall and during the index episodes will be reported.
Duration of Anti-CMV Therapy During CMV Episodes | Up to 7 years 3 months
  CMV episode is generally characterized by elevated CMV viremia levels resulting in anti-CMV treatment. Duration of anti-CMV therapy during CMV episodes will be reported.
Number of Participants With Distribution of Switches of Anti-CMV Agents at the Index Date | Up to years 3 months
  Index date is the date when participant was considered resistant, refractory or intolerant to anti-CMV treatment for the first time after transplant (RRI CMV index date) or pre-emptive treatment for the first time after transplant following CMV viremia (CMV preemptive treatment index date. Number of participants with distribution of switches of anti-CMV agents at the index date will be reported.
Percentage of Participants Administered With First, Second, Third and Fourth Line of Anti-CMV Treatments From HSCT | Up to 7 years 3 months
  Percentage of participants administered with first, second, third and fourth line of anti-CMV treatments from HSCT will be reported.
Time from HSCT to Administration of First-line Anti-CMV Agents of Interest and Between First-line Through the Fourth Line of Treatment | Up to 7 years 3 months
  Anti-CMV agents of interest includes specifically ganciclovir, valganciclovir, foscarnet, cidofovir, letermovir and maribavir, ganciclovir and foscarnet, valganciclovir and foscarnet, cidofovir and valganciclovir, cidofovir and valganciclovir, others which includes acyclovir, valacyclovir, immunoglobulin G (IgG), etc.
Number of Participants Based on Reasons for Anti-CMV Dose Changes or Discontinuation for Anti-CMV Agents of Interest | Up to 7 years 3 months
  Recurrent episodes is defined as new CMV infection in a participant with previous evidence of CMV infection. Index episode is first CMV episode in which the participant is considered RRI to anti-CMV treatment or had CMV viremia and received pre-emptive treatment, without becoming RRI during that episode. CMV episode is generally characterized by elevated CMV viremia levels resulting in anti-CMV treatment. Number of participants based on reasons for anti-CMV dose changes or discontinuation for anti-CMV agents of interest overall during CMV episodes, the index episode and for recurrent episodes will be reported.
Number of Participants With Anti-CMV Agent Administered When Diagnosed With Myelosuppression and Nephrotoxicity | Up to 7 years 3 months
  Index episode is first CMV episode in which the participant is considered RRI to anti-CMV treatment or had CMV viremia and received pre-emptive treatment, without becoming RRI during that episode. CMV episode is generally characterized by elevated CMV viremia levels resulting in anti-CMV treatment. Number of participants with anti-CMV agent administered when diagnosed with myelosuppression and nephrotoxicity at the index episode and during CMV episodes overall will be reported.
Number of Participants Using Immunosuppressant From HSCT | Up to 7 years 3 months
  Number of participants using immunosuppressant from HSCT will be reported.
Number of Participants With CMV-related Outpatient Clinic Visits From HSCT and Index Date | Up to 7 years 3 months
  Index date is the date when participant was considered resistant, refractory or intolerant to anti-CMV treatment for the first time after transplant (RRI CMV index date) or pre-emptive treatment for the first time after transplant following CMV viremia (CMV preemptive treatment index date. Number of CMV-related outpatient clinic visits from HSCT and index date will be reported.
Number of Participants Based on Selected Procedures Performed at Outpatient Clinical Visits From HSCT and Index Date | Up to 7 years 3 months
  Index date is the date when participant was considered resistant, refractory or intolerant to anti-CMV treatment for the first time after transplant (RRI CMV index date) or pre-emptive treatment for the first time after transplant following CMV viremia (CMV preemptive treatment index date. Selected procedures include preemptive monitoring, diagnostic imaging, treatment infusion, toxicities from anti-CMV agents.
Number of Participants Based on CMV-related Hospitalizations and Emergency Department Visits From HSCT and Index Date | Up to 7 years 3 months
  Index date is the date when participant was considered resistant, refractory or intolerant to anti-CMV treatment for the first time after transplant (RRI CMV index date) or pre-emptive treatment for the first time after transplant following CMV viremia (CMV preemptive treatment index date. Number of participants based on CMV-related hospitalizations and emergency department visits from HSCT and from index date will be reported.
Number of Participants Categorized Based on Reasons for CMV-related Hospitalization | Up to 7 years 3 months
  Primary reason for hospitalization will include treatment infusions, CMV progression. Number of participants categorized based on reasons for CMV-related hospitalization will be reported.
Number of Participants Based on Selected Procedures Performed at Hospitalizations and Emergency Department Visits From HSCT and Index Date | Up to 7 years 3 months
  Index date is the date when participant was considered resistant, refractory or intolerant to anti-CMV treatment for the first time after transplant (RRI CMV index date) or pre-emptive treatment for the first time after transplant following CMV viremia (CMV preemptive treatment index date. Selected procedures will include diagnostic imaging, treatment infusion, toxicities from anti-CMV agents.
Length of Hospital Stay for CMV-related Hospitalizations and Hospital Acquired CMV Viremia | Up to 7 years 3 months
  Length of hospital stay in days for CMV-related hospitalizations and hospital acquired CMV viremia will be reported.
Duration of Stay in Critical Care and Non-critical Care | Up to 7 years 3 months
  Duration in days of stay in critical care and non-critical care will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (11):
- MU Graz, Graz, Austria
- UZ Leuven, Leuven, Belgium
- Canada (2):
  - Hamilton Health Sciences Corporation, Hamilton, Ontario
  - McGill University Health Centre, Montreal, Quebec
- Greece (2):
  - Attikon General University Hospital, Athens
  - George Papanikolau, Thessaloniki
- Israel (2):
  - Rambam Health Care Campus, Haifa
  - Chaim Sheba Medical Center, Ramat Gan
- Institute of Hematology and Transfusion Medicine (IHTM), Warsaw, Poland
- Serbia (2):
  - University Clinical Center of Serbia, Belgrade
  - Clinical Center of Vojvodina, Novi Sad

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/ebaa078d48c24d93?idFilter=%5B%22TAK-620-4004%22%5D